CLINICAL TRIAL: NCT03453606
Title: Respiratory Rehabilitation at Home vs in the Center for Patients With Chronic Obstructive Pulmonary Disease: Efficacy, Preferences and Costs
Brief Title: Respiratory Rehabilitation for Patients With Chronic Obstructive Pulmonary Disease
Acronym: REHABDO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of inclusion
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017_08; 2017-A02393-50 (Other: ID-RCB number, ANSM); PREPS-16-249 (Other: PREPS number, DGOS)
Record Dates: First submitted 2018-02-16; First posted 2018-03-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary rehabilitation; home-based
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home group (Active Comparator)
  Interventions: Other: Home respiratory rehabilitation
- center group (Active Comparator)
  Interventions: Other: Center respiratory rehabilitation

INTERVENTIONS:
Other: Home respiratory rehabilitation — Home care is individual (often with the spouse or the carer), during 1h30, one visit per week for 8 weeks, after completion of the educational diagnosis, under direct supervision of a member of the team, with continued physical activities in autonomy the others days of the week, according to a personalized action plan. No visit is scheduled in the pulmonologist, the general practitioner or in the rehabilitation center. The team includes pulmonologist, nurses, dietician, socio-medical beautician and a administrative assistant.
  Arms: home group
Other: Center respiratory rehabilitation — In an outpatient setting, the course is performed in groups of 6 to 8 patients, during sessions from 3 to 7 am, under the direction of health professionals, 3 to 5 times a week, for 4 to 6 weeks, for a total of 20 to 24 sessions. Internally, patients come to "complete" hospitalization for 4 weeks. This duration can be modulated according to the evolution of the patients.
  Supervision is carried out by the entire team including pulmonologists, nurses, physiotherapists, psychologists, activity professors adapted physicists, dietician
  Arms: center group

SUMMARY:
The aim of this clinical trial is to establish the non-inferiority of home-based respiratory rehabilitation compared to respiratory rehabilitation in center in terms of exercise tolerance as evaluated by the 6 minutes Stepper test..

This trial will also 1°) evaluate the Medico-economic aspects of the home-based Respiratory rehabilitation versus respiratory Rehabilitation in center; 2°) analyse the patient preferences between home-based respiratory rehabilitation and respiratory rehabilitation in center and 3°) Compare home-based respiratory rehabilitation vs respiratory rehabilitation in center in terms of dyspnea, quality of life, anxiety and depression.

DETAILED DESCRIPTION:
The purpose of this study is to perform a comparative analysis of the clinical and medico-economic effectiveness of center-based RR versus home-based RR in the departments of Nord and Pas de Calais in France. All COPD patients eligible for RR and willing to participate in the study will be followed.

Patient preferences will be evaluated at inclusion. After presentation of both RR modalities, patients expressing a strong preference for one or other of the terms will be taken care of according to their wishes. Indifferent patients between the two RR modalities will be randomized.

This design is justified in the light of three cases:

* It is impossible to evaluate blind intervention,
* The effectiveness of RR depends on patient preferences,
* Patients' adherence to the protocol is facilitated.

ELIGIBILITY:
Inclusion Criteria:According to HAS recommendations, SPLF, ERS / ATS (3) (18) (19) can be included any patient, over 18 years old, with stage II - III - IV COPD presenting disabling dyspnoea in activities of daily living, and / or in the course of acute exacerbation of COPD (EABPCO), with no other respiratory pathology diagnosed.

Exclusion Criteria:

According to the recommendations, HAS, SPLF, ERS / ATS will not be included any patient having :

* co-morbidities including unstabilized cardiovascular disease,
* significant cognitive disorders: patients with a history of pathologies neurodegenerative with loss of mental faculties (example: Alzheimer)
* psychiatric disorders: patients with impaired judgment and perception
* neurological or orthopedic disorders that do not allow the realization of physical activities

Also, will not be included, the patient (s):

* waiting for lung transplantation,
* pregnant or nursing,
* in an emergency situation
* unable to receive enlightened information,
* unable to participate in the entire study,
* not covered by the social security scheme,
* refusing to sign the consent,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline the 6 minutes Stepper test at 2 months | At 2 months
  The 6 minutes stepper test (ST6), performed on a Stepper allows to analyze the number of strokes (or steps) performed in 6 minutes

SECONDARY OUTCOMES:
Change from baseline the 6 minutes Stepper test at 6 and 12 months | at 6 months, at12 months
  The 6 minutes stepper test (ST6), performed on a Stepper allows to analyze the number of strokes (or steps) performed in 6 minutes
Percentage of patients expressing a preference marked for home-based respiratory rehabilitation or respiratory rehabilitation in center | Baseline
Cost of interventions: respiratory rehabilitation in center or at home | At 12 months
Change from Baseline COPD Assessment Test (CAT) at 2,6,12 months | baseline, after RR (2 months); 6 months and12 months
  The COPD assessment test (CAT) is a short questionnaire initially intended for assess quality of life and clinical impact of COPD
Change from Baseline Modified Medical Research Council (MMRC) Dyspnea Scale at 2,6,12 months | baseline, after RR (2 months); 6 months and12 months
  The scale measures a person's limitation base on a scale of 0-4 and uses the final value to determine how much disability is caused by shortness of breath.Five-option grading system called the Modified Medical Research Council (MMRC) Dyspnea Scale.
Change from Baseline Anxiety and Depression (HAD) at 2,6,12 months | Baseline, after RR (2 months); 6 months and12 months
  To determine the levels of anxiety and depression that a COPD patients are experiencing
EPICES score | baseline
  EPICES score (Assessment of the precariousness and health inequalities in the Health Examination Centers, French) is an individual indicator of precariousness
  ,Self-administered questionnaire,quantify the level of social vulnerability and precariousness. It ranges from zero (no vulnerability) to 100 (maximum vunerability)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Le Rouzic, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - Centre hospitalier de béthune, Béthune
  - CH de Béthune, Béthune
  - Hôpital Calmette, CHU, Lille
  - CH de Loos, Loos
  - CH Victor Provot, Roubaix, Roubaix
  - CH de Tourcoing, Tourcoing
  - CH de Wattrelos, Wattrelos